CLINICAL TRIAL: NCT05933876
Title: Stereotactic ABlative Radiotherapy (SABR) in Oligometastatic Cancer (OC): a Radiomics, Multi-omics, and Machine Learning Approach to Clinical Decision-making. the OC-SABR Multicentric Project
Brief Title: The Impact of Radiotherapy on Oligometastatic Cancer
Status: Recruiting | Type: Observational
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: Hospital Ruber Internacional (Other); Hospital Universitario Rey Juan Carlos (Other); Quirón Madrid University Hospital (Other); Hospital de La Luz (Other); Institut Català d'Oncologia (Other); Hospital Arnau de Vilanova (Other); Hospital Universitari Sant Joan de Reus (Other); Hospital Universitario Virgen Macarena (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospital General Universitario de Valencia (Other); Hospital Clínico Universitario de Valencia (Other); Complejo Hospitalario Universitario de Albacete (Other); Hospital de Terrassa (Other); Hospital Universitario Ramon y Cajal (Other); Hospital del Mar (Other); Hospital Provincial de Castellon (Other); Hospital de la Santa creu i Sant Pau - Barcelona (Other); HM Sanchinarro University Hospital (Other); Hospital Miguel Servet (Other); University Hospital Virgen de las Nieves (Other); Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Other Study IDs: OC-SABR
Record Dates: First submitted 2023-03-28; First posted 2023-07-06 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Metastasis; Metastatic Breast Cancer; Metastatic Prostate Cancer; Metastatic Colorectal Cancer; Metastatic Lung Cancer
Keywords: Metastasis; Radiosurgery; Metabolomics; Radiomics; Multi-omics; Molecular subtypes
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Plasma, serum, and DNA samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OC-SABR: Patients diagnosed with Oligometastatic Cancer (OC) that will receive Stereotactic ABlative Radiotherapy (SABR) that has been prescribed per clinical protocol.
  Interventions: Diagnostic Test: To propose a diagnostic test to determine the viability of Stereotactic ABlative Radiotherapy (SABR).; Diagnostic Test: To propose a diagnostic test to determine the effectiveness of SABR.; Diagnostic Test: To propose a diagnostic test for Oligometastatic Cancer (OC).
- Controls: Individuals who have never been diagnosed with cancer or oligometastasis.
  Interventions: Diagnostic Test: To propose a diagnostic test for Oligometastatic Cancer (OC).

INTERVENTIONS:
Diagnostic Test: To propose a diagnostic test to determine the viability of Stereotactic ABlative Radiotherapy (SABR). — Analyze clinical data, medical images and molecular circulating features to propose which variables serve to select the patients that will achieve complete response after SABR.
  Groups: OC-SABR
Diagnostic Test: To propose a diagnostic test to determine the effectiveness of SABR. — Collect blood samples at five different time points before and after treatment and analyze circulating tumoral DNA, medical images, and metabolites to monitor the effect of SABR and its effectiveness.
  Groups: OC-SABR
Diagnostic Test: To propose a diagnostic test for Oligometastatic Cancer (OC). — Analyze circulating tumoral DNA and metabolites from blood samples in search of the profile of OC.

SUMMARY:
Metastases represent the most threatening challenge in cancer. One of the management strategies for patients with Oligometastatic Cancer (OC) is Stereotactic ABlative Radiotherapy (SABR). However, there are few studies, and there is no defined clinical standard, nor are the radiobiological mechanisms that contribute to treatment response well understood. The focus should be on generating evidence to guide the personalization of radiotherapy beyond solely technological and anatomical precision. This could be achieved by recollecting clinical and biological data from patients that undergo this treatment and analyzing them to ultimately predict, with the help of artificial intelligence, which patients will be the most beneficiary and improve their survival rate.

DETAILED DESCRIPTION:
Metastases are the most threatening challenge in cancer. In patients with metastatic cancer, local radiotherapy treatment remains an essential tool with different goals that depend on numerous factors, especially on the number and extent of the metastases and whether disease control is feasible and desirable according to the expected quality of life. Oligometastatic Cancer (OC), i.e., a few metastases in a few organs, has been recently incorporated as a less aggressive state than widely disseminated metastatic disease. Consequently, OC is a serious candidate for aggressive treatments based on Stereotactic ABlative Radiotherapy (SABR). This treatment has shown promising results and is already incorporated into habitual clinical practices. However, OC is a complex and heterogeneous disease, and not all patients have improved their life quality and expectation. Identifying patients who would benefit from this treatment is an important area of research that needs factual information from a large sample provided by multiple centers. Therefore, this multicenter, retrospective, prospective, observational, and longitudinal study incorporates clinical data, medical images, and biological samples to feed artificial intelligence algorithms. The objective is to determine which patient profile achieves complete response after SABR. The secondary objectives are:

1. To analyze metastases by radiomics using computed tomography, magnetic resonance, or positron emission tomography images; and
2. To evaluate intratumoral metabolites released into circulation by multi-omics analyses.

These will contribute to determining the systemic molecular effects of treatment in search of biomarkers with predictive value.

Centralized storage of patient management data, clinical image analysis, and candidate biomarkers measured in blood samples may eventually meet the expectations of integrating data into clinical decision-making and influence evolution based on precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of primary tumor: breast, prostate, lung, colorectal.
* 18 years old or older.
* Up to five metastases located in the bone, lung, node, liver or brain.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Scale 0 or 1.

Exclusion Criteria:

* Non-melanoma skin cancer.
* Previous radiotherapy in the same anatomic location.
* Presence of vascular collagen disease.
* Pregnancy or lactation at the time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the collaboration hospitals to receive Stereotactic ABlative Radiotherapy (SABR) to treat Oligometastatic Cancer (OC).
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2037-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiological rate | 3 months after treatment
  Images obtained by computerized tomography, magnetic resonance and positron emission tomography serve to evaluate the local control and response rate by:
  * Complete response: absence of disease.
  * Stable disease: no changes.
  * Partial response: 50% or more injury reduction.
  * Progression: 25% or more tumor size increase.
  According to RECIST Criteria 1.1 and PERCIST.
Progression-Free Survival | 5 years after treatment
  To assess the impact of SABR on the progression over time, precisely at 1, 2, 3, and 5 years, regarding Progression-Free Survival (PFS) based on RECIST Criteria 1.1 and PERCIST.
SABR toxicities | 5 years after treatment
  To evaluate the progression of SABR toxicities over time, precisely at 1, 2, 3, and 5 years, according to the CTCAE 4.0 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Meritxell Arenas, PhD., Study Director — Universitat Rovira i Virgili, Hospital Universitari Sant Joan de Reus
Locations (21):
- Spain (21):
  - Complejo Hospitalario Universitario Albacete, Albacete, Albacete
  - Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Institut Català d'Oncologia, Barcelona, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Universitari Arnau de Vilanova, Lleida, Lleida
  - Hospital de La Luz, Madrid, Madrid
  - Hospital Ruber Internacional, Madrid, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid, Madrid
  - Hospital Universitario Quirónsalud, Madrid, Madrid
  - Hospital Universitario Rey Juan Carlos, Madrid, Madrid
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital General Univesitario de Valencia, Valencia, Valencia
  - Hospital Universitari Miguel Servet, Zaragoza, Zaragoza
  - Hospital del Mar, Barcelona
  - Hospital Provincial de Castellón, Castellon
  - Institut Català d'Oncologia, Girona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital de Terrassa, Terrassa

IPD SHARING:
Plan to Share IPD: Yes
The Data Management Plan makes data fully findable, accessible, interoperable, and reusable, following the indication of the Horizon 2024 initiative of the European Union. The clinical team identified sensitive data, including epidemiological, anthropometric, and medical information. It is the only responsibility of the principal investigator to ensure that sensitive data are de-identified, implementing technical safeguards to guarantee anonymity.
  Most data will be experimental and obtained from the analysis of column value and data format description (.txt or .csv) and syntax scripts (.R).
  The external collaborators, especially those involved in validation cohorts, may have access to data upon request.
  With the acceptance of the principal investigator, Rovira i Virgili University's institutional service will guarantee digital access to repositories with raw data generated in research analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Once decided the repository web address.
Access Criteria: Decided by the principal investigator.